CLINICAL TRIAL: NCT05792592
Title: Small Airways Disease (SAD) in Severe Asthma as a Novel Endpoint and Distinct Target for Biological Therapy. Small Airways Disease (SAD) in Severe Asthma as a Novel Endpoint and Distinct Target for Biological Therapy (SASAB Study)
Brief Title: Small Airways Disease (SAD) in Severe Asthma as a Novel Endpoint and Distinct Target for Biological Therapy.
Acronym: SASAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, BONINI MATTEO, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4253
Record Dates: First submitted 2023-03-07; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Small Airway Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uncontrolled Severe asthmatics: Uncontrolled Severe asthmatics
  Interventions: Diagnostic Test: IOS (Impulse Oscillometry)

INTERVENTIONS:
Diagnostic Test: IOS (Impulse Oscillometry) — Small Airways Disease Assessment

SUMMARY:
Severe asthma is now widely accepted to be a heterogeneous syndrome consisting of multiple phenotypes identified by specific biomarkers and targeted by tailored biological therapies. However, much remains unclear regarding the best approaches to manage these patients, or concerning the pathophysiological mechanisms underlying the disease.

Small airway (SA) are defined as those airways with an internal diameter <2 mm. In patients affected by asthma, it has been reported that SA are the predominant site of airflow resistance. Peripheral airways are thickened in asthma due to chronic inflammation in the epithelium, submucosa and muscle area. It has been suggested that the outer wall is more inflamed than the inner wall, with a higher number of lymphocytes, eosinophils, and neutrophils associated to an increased expression of interleukin-4 (IL-4), interleukin-5 (IL-5) and eotaxin. Moreover, it is well documented that SA inflammation and dysfunction contribute significantly to the clinical impact of asthma and that 50-60% of asthmatics have a SA involvement across all disease severities. An important question is whether SA disease in asthma is variable among distinct asthma phenotypes and whether it occurs in all patients. Cluster analyses have been recently used to identify specific asthma phenotypes, but markers of SA function have not been investigated. However, evidence is accumulating to support that SA dysfunction and inflammation may contribute to distinct asthma phenotypes. Recent findings indicate that SA are significantly affected in severe asthma and that their involvement is associated with worse disease outcomes. It has been reported that patients with asthma and a history of frequent exacerbations per year had a significant SA involvement. Furthermore, peripheral airways significantly contribute not only to the level of asthma control, but also to patients' quality of life and perception of symptoms. At last more thickened SA and higher numbers of eosinophils are detectable in subjects with fatal asthma.

The assessment of SA represents a big challenge and requires qualified expertise and sophisticated techniques including body plethysmography, single and multiple breath nitrogen washout, impulse oscillometry (IOS), fraction exhaled NO at multiflow, sputum induction and high-resolution chest CT (HRCT). Such procedures can either provide functional information on the degree/extent of ventilation heterogeneity and air trapping or facilitate the understanding of the inflammatory and remodeling processes.

In addition, a number of clinical trials have in recent years demonstrated the efficacy of biologics in severe asthma. Omalizumab, a humanized anti-Imunoglobulin E monoclonal antibody (mAb) has been well recognized as an important option for treating allergic asthma as an add- on therapy for uncontrolled disease.

Three anti-IL-5 therapies are currently available for the treatment of severe asthma, including Mepolizumab, Reslizumab, and Benralizumab.

The newest biologic agent to be approved is Dupilumab that is a human mAb that targets the subunit of the IL-4 receptor.

Biologics represent an innovative strategy for the treatment of severe asthma. In most patients with SAD these drugs control inflammation, improve lung function, ameliorate clinical symptoms, reduce exacerbations and have a marked steroid-sparing effect. However, there is still a significant proportion of non-responders and a lack of validated predictive biomarkers in such subpopulation. In regard to this, very limited findings are available about the effect of biologics therapy on SA.

DETAILED DESCRIPTION:
Study hypothesis We hypothesize that biological therapy has a significant beneficial effect on small airways disease in severe asthmatics and that the evaluation of small airways before and during treatment may represent a distinctive marker of response and a novel target for a preferential use of one over other biological therapies currently available for severe asthmatic patients.

Study objectives

* To evaluate small airway endpoints in severe asthmatics before starting biologic treatment.
* To evaluate longitudinal changes of these endpoints at different time points during biologic treatment.
* To relate small airway endpoints recorded at baseline and their changes over time to other functional, laboratory, clinical and patient-reported outcomes.
* To make comparisons for subgroups identified on the basis of the type of the biological drug used.

Study center

The study will be conducted at the Asthma Center of Fondazione Policlinico Universitario Agostino Gemelli. Asthma Clinic evaluates approximately 1000 asthmatic patients per year; furthermore, it is part of the Italian Severe Asthma Network (SANI) and one of the coordinating centers for the newborn Italian Mild-Moderate Asthma Network (MANI), therefore representing a center of excellence and reference at a national level, with easy and wide access to the study population.

Study design This is a 24-month, single-site observational retrospective and prospective longitudinal cohort study involving asthmatic patients referred to the Asthma Center and eligible for starting one of the biological therapy currently available. The patient will be considered eligible only after having optimized adherence, inhalation technique, comorbidity management and following a multidisciplinary assessment. Subjects will be monitored for 12 months and SA endpoints as well as other functional, clinical, laboratory and patient-reported outcomes will be recorded at the beginning of the biological therapy (T0) and after 3,6,12 months (T3, T6, T12). Values and changes in SA endpoints will be also related to other functional, clinical and patient-reported outcomes.

Study procedures

The following study procedures will be performed in the framework of the standard care for severe asthmatic patients:

* Clinical history;
* Demographics data (such as age, sex, race et.)
* Questionnaires (i.e. Asthma Control Test [ACT], Asthma Control Questionnaire [ACQ], Asthma Quality of Life Questionnaire [AQLQ])
* Pulmonary function tests (i.e. spirometry [Forced Expiratory volume in 1 second (FEV1),Forced Vital Capacity (FVC), FEV1/FVC, body plethysmography [Residual Volume (RV), Total Lung Capacity (TLC), RV/TLC, impulse oscillometry as resistance at 5 and 20 Hz (R5, R20).
* Airway inflammatory markers (i.e. fraction exhaled nitric oxide - FeNO)
* Allergy tests (i.e. skin-prick tests and immunoassays for total and specific serum IgE)
* Biological sampling (i.e. blood and sputum eosinophils).
* Imaging (i.e. chest XR and HRCT)

Study endpoints The primary endpoint will be represented by the R5-R20 parameter registered through impulsoscillometry. Baseline values and changes over the one-year follow-up period at preplanned timepoints (i.e. 3, 6, and 12 months) will be recorded. According to literature evidence, baseline values ≥0.07 support the evidence of small airways dysfunction.

Secondary endpoints will be represented by indirect parameters of SA involvement (i.e. TLC, RV, TLC/RV, FEF25-75). Baseline values and changes over the one-year follow-up period at preplanned timepoints (i.e. 3, 6, and 12 months) will be recorded.

Variations in primary and secondary endpoints will be also related to changes in functional parameters (i.e FEV1), clinical parameters (exacerbation rate), inflammatory markers (FeNO) and patients' questionnaire scores (ACT, AQLQ, ACQ). Established minimal clinically important difference (MCID) thresholds will be taken into consideration for correlation analyses.

Statistical analysis Statistical analysis will be performed using a statistical software. Data will be tested for normality and will be expressed as mean (SD) or median (IQR). Comparative analysis will be performed using parametric and non-parametric methods as appropriate. Single and multiple linear regression analyses will be run to determine correlation between small airway endpoints and clinical, functional, laboratory, and patients' reported outcomes. A p-value≥0.05 will be considered statistically significant. Most appropriate statistical analyses and models will be anyway chosen and run, following the advice of statisticians at the institutional Department of Public Health. Considering the "R5-R20 Delta", measured through impulse oscillometry, as the primary endpoint for the study, and aiming for a minimal difference of 0.02 (according to literature data), in order to have an a error of 0.5 and a study power of 80%, at least 54 subjects will have to be enrolled in the study. Documentation will be stored for a minimum of 10 years after the completion of the study, including the follow-up period.

Study significance and innovation Systems biology approaches are establishing the links between disease pathways/mechanisms, and clinical/physiologic features. Validation of these pathways may contribute to better defining severe asthma endotypes and treatable mechanisms. Precision medicine approaches are necessary to link treatable mechanisms with treatable traits and biomarkers derived from clinical, physiologic, inflammatory, molecular and genetic variables. A deep and proper assessment of airway samples along with non-invasive biomarkers may have a highly relevant translational significance and enable better knowledge and management of severe asthma.

Risk analysis No major difficulties are expected in view of the study's observational design. No additional costs will be held.

ELIGIBILITY:
* Adult (≥ 18 years) male and female subjects,
* Capable to sign the informed consent,
* Severe asthma (≥12months high-dose inhaled corticosteroids + additional controller treatments) and ≥ 2 exacerbations (corticosteroid and/or Emergency Department visit and/or hospitalization in the previous 12 months);
* eligible for the administration of one of the approved biological therapy currently available.
* A smoking history <2 pack/year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥ 18 years) male and female subjects, capable to sign the informed consent, addressed to the Asthma Center, with severe asthma as defined by current guidelines (≥12months high-dose inhaled corticosteroids + additional controller treatments) and ≥ 2 exacerbations (corticosteroid and/or Emergency Department visit and/or hospitalization in the previous 12 months). The patient should have a smoking history <2 pack/year and should be eligible for the administration of one of the approved biological therapy currently available.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2024-06-16 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline of R5-R20 over one-year follow-up after the beginning of biological therapy | Baseline, and after 3, 6 and 12 months.
  R5-R20

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bonini, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No